CLINICAL TRIAL: NCT01494662
Title: A Phase II Trial of HKI-272 (Neratinib), Neratinib and Capecitabine, and Ado-Trastuzumab Emtansine for Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer and Brain Metastases
Brief Title: HKI-272 for HER2-Positive Breast Cancer and Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Puma Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-344; TBCRC 022 (Other: TBCRC)
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Results first posted 2024-05-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: HER2 Positive; BrCa
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Biopsy; Capecitabine; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Active Comparator): Patients With Progressive Brain Metastases
  Intervention: HKI-272 (Neratinib)340 mg orally, once daily.
  Interventions: Drug: HKI-272
- Cohort 2 (Active Comparator): Patients Who Are Candidates For Craniotomy.
  Intervention: HKI-272 (Neratinib) 240 mg orally, once daily.
  Surgical resection (biopsy).
  Neratinib concentrations from craniotomy specimen, CSF, plasma Neratinib.
  Interventions: Procedure: Surgical Resection
- Cohort 3a/3b (Active Comparator): Cohort 3a will be made up of participants with No Prior Lapatinib Treatment. They will receive Neratinib 240mg Orally daily and 750mg/m2 Capecitabine twice per day for 14 days followed by 7 days rest.
  Cohort 3b will be made of of participants with Prior Lapatinib Treatment. Cohort 3b participants will receive Neratinib 240mg Orally daily and 750mg/m2 Capecitabine twice per day for 14 days followed by 7 days rest.
  Interventions: Drug: Capecitabine
- Cohort 4a/4b/4c (Active Comparator): Cohort 4a will be made up of participants with previously untreated brain metastases. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
  Cohort 4b will be made up of participants with progressive brain metastases. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
  Cohort 4c will be made up of participants with progressive brain metastases and prior T-DM1. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
  Interventions: Drug: HKI-272; Drug: Ado-Trastuzumab Emtansine

INTERVENTIONS:
Drug: HKI-272 — 240 mg orally, once daily
  Other Names: Neratinib
  Arms: Cohort 1
Procedure: Surgical Resection — Neratinib concentrations from craniotomy specimen, CSF, plasma Neratinib.
  Other Names: Biopsy
  Arms: Cohort 2
Drug: Capecitabine — 750 mg/m2 orally, twice daily (1,500 mg/m2 daily) for 14 days followed by 7 days off
  Other Names: Xeloda
  Arms: Cohort 3a/3b
Drug: HKI-272 — 160 mg orally, once daily
  Other Names: Neratinib
  Arms: Cohort 4a/4b/4c
Drug: Ado-Trastuzumab Emtansine — 3.6 mg/kg IV every 3 weeks
  Other Names: T-DM1
  Arms: Cohort 4a/4b/4c

SUMMARY:
The purpose of this research study is to determine how well neratinib works in treating breast cancer that has spread to the brain. Neratinib is a recently discovered oral drug that may stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2).

In this research study, the investigators are looking to see how well neratinib works to decrease the size of or stabilize breast cancer that has spread to the brain. The investigators are also looking at how previous treatments have affected your thinking (or cognition) and how much neratinib reaches the central nervous system.

DETAILED DESCRIPTION:
Subjects will receive neratinib and a drug-dosing calendar for each treatment cycle. This drug is given orally on a daily basis, continuously. Each treatment cycle will last for 4 weeks during which time the subject will be taking neratinib every day.

* Physical Exams and vital signs: At the start of each cycle, you will have a physical exam. You will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. You will also have a neurological examination to assess for neurological symptoms.
* Scans (or Imaging tests): We will assess your tumor by brain MRI every 2 cycles ( 6 to 8 weeks) and then every 3 cycles (9 to 12 weeks). CT or MRI scans of your chest, abdomen, and pelvis will be performed every other cycle, at the same time points as the brain MRI. Your research doctor may ask you to have a bone scan at the same time points if this is clinically indicated.
* Photographs: Photographs may be taken of your tumor to assess the response of your tumor to the treatment. Care will be taken to ensure these do not reveal your identity.
* MUGA or Echo: You will have a MUGA or ECHO done every 12 weeks, so every 3 or 4 treatment cycles, depending on which cohort you are on.
* Blood tests: You will have blood tests done at the beginning of each treatment cycle to check your blood cell counts and how well your organs are functioning. In addition to regular blood tests, we will be collecting 2-3 tablespoons of blood for research prior to your study treatment start.
* Neurocognitive Function: If you have previously received treatment for cancer that has spread to your brain (prior to enrollment on this study), you will be asked to take a battery of tests that assess your cognition (thinking) at the start of the study, after 2 cycles of treatment, and possibly at the end of the study. With these tests, we are trying to better understand how your previous treatments and ongoing treatments affect your memory, attention, learning, and other related skills. These tests will be administered to you by a trained research assistant and may take 30-45 minutes to complete.
* For preoperative patients only: If you are a patient who is planning to have an operation to remove the cancer in your brain, you will have your surgery between 7-21 days after starting neratinib. These tests will allow us to measure of how much drug (neratinib) reaches the central nervous system and will help us understand how well neratinib does this.
* At surgery, a part of your tumor cerebrospinal fluid will be collected to test for levels of neratinib. For the cerebrospinal fluid collection, this may require a lumbar puncture just before your surgery begins (spinal tap) if your neurosurgeon feels he/she cannot collect this fluid easily during your surgery. A lumbar puncture is a test often used to detect tumor cells in your cerebrospinal fluid. In this case, we will collect fluid for testing of cancer cells and will also examine the fluid for neratinib concentrations. This will provide information on how much drug (neratinib) reaches the central nervous system. There will be a separate consent form for this procedure given to you by your neurosurgeon (when applicable). This procedure will be done while you are already under general anesthesia for your surgery. If you have a contraindication to having this procedure or if you wish to refuse to undergo this procedure, you may do so.
* You will also have a blood test on day of surgery to test for levels of neratinib
* You will then resume neratinib once you have recovered from your surgery

After the final dose of the study drug:

You will have a follow-up visit one month after coming off study treatment. During that visit, you will have a physical examination, functional assessment, assessment of any toxicities and current medications, and a neurological examination. If you continue to have ongoing toxicity related to your study treatment, we will continue to follow you until this toxicity resolves. In addition, we will collect about 5-6 tablespoons of blood for research and to measure if a marker for your particular breast cancer exists.

We would like to keep track of your medical condition for up to two years after you stop the study treatment. If you are not seen in follow-up at your participating center (where you enrolled on the study), we would like to follow you by calling you on the telephone or by sending you a letter once a year to see how you are doing. We may also contact your doctor once every 6 months to see how you are doing. Keeping in touch with you and checking your condition every year helps us look at the long-term effects of the research study. If you do not wish to be contacted after you stop the study treatment, you must notify the research study staff of your withdrawal of consent for follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients (men or women) must have histologically or cytologically confirmed invasive breast cancer, with metastatic disease. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis by physical exam or radiologic study.
* Invasive primary tumor or metastatic tissue confirmation of HER2-positive status
* Over-expression by immunohistochemistry (IHC) with score of 3+ (in > 30% of invasive tumor cells) AND/OR HER2 gene amplification (> 6 HER2 gene copies per nucleus or a FISH ratio [HER2 gene copies to chromosome 17 signals] of ≥ 2.0)
* Note: Patients with a negative or equivocal overall result (FISH ratio of < 2.0 or ≤ 6.0 HER2 gene copies per nucleus) and IHC staining scores of 0, 1+, 2+ are not eligible for enrollment
* No increase in corticosteroid dose in the week prior to baseline brain MRI
* Prior trastuzumab and lapatinib therapy are allowed.
* There is no limit to the number of previous lines of therapy (including chemotherapy, trastuzumab, and endocrine therapies)
* No prior therapy with neratinib is allowed
* At least 2 weeks washout period post chemotherapy, any prior protocol therapy, lapatinib, other targeted or biologic therapy, or radiation therapy is required prior to study entry
* No washout is required for hormonal therapy but concurrent hormonal therapy is not allowed for patients on study

Patients with progressive disease (Cohort 1):

* For cohort 1, patients must have new or progressive CNS lesions, as assessed by the patient's treating physician.
* In cohort 1, patients must have measurable CNS disease, defined as at least one parenchymal brain lesion that can be accurately measured in at least one dimension with longest dimension ≥10 mm by local radiology review. Note: measurable non-CNS disease is NOT required for study participation
* It is anticipated that some patients may have multiple progressive CNS lesions, one or several of which are treated with SRS or surgery with residual untreated lesions remaining. Such patients are eligible for enrollment on this study providing that at least one residual (i.e. non-SRS-treated or non-resected) lesion is measurable (≥10 mm).
* Patients who have had prior cranial surgery are eligible, provided that there is evidence of measurable residual or progressive lesions, and at least 2 weeks have passed since surgery. If a patient has surgical resection followed by WBRT, then there must be evidence of progressive CNS disease after the completion of WBRT.
* Patients who have had prior WBRT and/or SRS and then whose prior treated lesions have progressed thereafter are also eligible. In this case, lesions which have been treated with SRS may be considered as target lesions if there is unequivocal evidence, in the opinion of the treating physician, of progression.

Patients with with operable disease (Cohort 2):

* In cohort 2, eligible patients will include those who have CNS disease that is amenable for surgery (typically < 3 brain metastases and with planned resection by neurosurgery). These patients may include those who have received or not received previous treatment(s) for their CNS.
* It is anticipated that that patients who have intracranial disease amenable to surgery will have measurable CNS disease prior to study entry and to resection. However, this is not an eligibility requirement. Measurable disease is also not required to continue on protocol subsequent to surgical resection.
* For patients who undergo surgery, postoperative whole brain radiation therapy will not be allowed while patients are on study (concurrent neratinib and radiation therapy has not been studied and toxicity of this is unknown). Patients will require discontinuation of neratinib if radiation therapy will be administered.

Patient Cohort 3:

-In cohort 3, eligible patients must have measurable Central Nervous System disease. Cohort 3a will have participants with no prior lapatinib therapy. Cohort 3b will have had prior lapatinib therapy.

Exclusion Criteria:

* Not pregnant or breastfeeding
* Participants who have had chemotherapy or radiotherapy (including investigational agents) within 2 weeks prior to entering the study or those who have not recovered adequately from adverse events due to agents administered more than 4 weeks earlier (excluding alopecia). Washout from trastuzumab is not required.
* Participants who are currently receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to neratinib
* Concurrent use of enzyme-inducing antiepileptic drugs (EIAEDs), including phenytoin, carbamazepine, oxcarbazepine, fosphenytoin, phenobarbital, pentobarbital, or primidone
* Patients who are receiving any cancer-directed concurrent therapy, such as concurrent chemotherapy, radiotherapy, or hormonal therapy while on study. Concurrent treatment with bisphosphonates is allowed but should be started before the first dose of neratinib.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* More than two seizures over the last 4 weeks prior to study entry
* Patients with known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Those with leptomeningeal metastases as the only site of CNS disease
* Significant malabsorption syndrome or inability to tolerate oral medications
* Any predisposing chronic condition resulting in baseline grade 2 or higher diarrhea

Patient Cohort 4:

- In cohort 4, eligible patients must have measurable Central Nervous System disease. Cohort 4a will have participants with previously untreated brain metastases. Cohort 4b will have participants with progressive brain metastases. Cohort 4c will have participants will have progressive brain metastases and prior T-DM1

Exclusion Criteria:

* Participants who are currently receiving any other investigational agents.
* Participants who have had chemotherapy or radiotherapy (including investigational agents) within 2 weeks prior to entering the study or those who have not recovered adequately from adverse events due to agents administered more than 4 weeks earlier (excluding alopecia). Washout from trastuzumab or hormonal therapy is not required.
* History of severe allergic reactions or intolerability attributed to compounds of similar chemical or biologic composition to neratinib and T-DM1 for Cohorts 4A-4C Concurrent use of enzyme-inducing antiepileptic drugs (EIAEDs), including phenytoin, carbamazepine, oxcarbazepine, fosphenytoin, phenobarbital, pentobarbital, or primidone
* Patients who are receiving any cancer-directed concurrent therapy, such as concurrent chemotherapy, radiotherapy, or hormonal therapy while on study. Concurrent treatment with bisphosphonates and denosumab is allowed for bony metastases but should be started before the first dose of neratinib.
* Any prior treatment with T-DM1 for Cohorts 4A-4B.
* For Cohorts 4A, 4B, and 4C: Patients with myocardial infarction or cardiomyopathy onset within the last 6 months are excluded
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Active hepatitis B or hepatitis C with abnormal liver function tests
* Active liver disease from autoimmune disorders or sclerosing cholangitis
* Lung disease from etiology other than metastatic breast cancer resulting in dyspnea at rest (4A-4C)
* More than two seizures over the last 4 weeks prior to study entry
* Patients with known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body. However, Head CT with contrast is allowed in place of MRI at baseline and throughout the study if MRI is contraindicated and a participant's CNS lesions are clearly measurable on the head CT.
* Those with leptomeningeal metastases as the only site of CNS disease
* Significant malabsorption syndrome or inability to tolerate oral medications
* Any predisposing chronic condition resulting in baseline grade 2 or higher diarrhea
* Inability to comply with study and/or follow-up procedures
* Individuals with a history of a different active malignancy are ineligible.
* Pregnant women are excluded from this study because neratinib (and other agents on study) is an agent with the potential for teratogenic or abortifacient effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, M.D., M.P.H., Principal Investigator — Dana-Farber Cancer Institute
Locations (18):
- United States (18):
  - University of California, San Francisco Medical Center, San Francisco, California
  - MedStar Georgetown Univeristy Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hosptial, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina at Chapel Hill - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UPMC Passavant Cranberry, Cranberry Township, Pennsylvania
  - Arnold Palmer Cancer Center-Greensburg, Greensburg, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Ortenzio Cancer Center, Mechanicsburg, Pennsylvania
  - UPMC Cancer Centers - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine Lester and Sue Smith Breast Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freedman RA, Gelman RS, Agar NYR, Santagata S, Randall EC, Gimenez-Cassina Lopez B, Connolly RM, Dunn IF, Van Poznak CH, Anders CK, Melisko ME, Silvestri K, Cotter CM, Componeschi KP, Marte JM, Moy B, Blackwell KL, Puhalla SL, Ibrahim N, Moynihan TJ, Nangia J, Tung N, Burns R, Rimawi MF, Krop IE, Wolff AC, Winer EP, Lin NU; Translational Breast Cancer Research Consortium (TBCRC). Pre- and Postoperative Neratinib for HER2-Positive Breast Cancer Brain Metastases: Translational Breast Cancer Research Consortium 022. Clin Breast Cancer. 2020 Apr;20(2):145-151.e2. doi: 10.1016/j.clbc.2019.07.011. Epub 2019 Aug 22. PMID 31558424
- [Derived] Freedman RA, Gelman RS, Anders CK, Melisko ME, Parsons HA, Cropp AM, Silvestri K, Cotter CM, Componeschi KP, Marte JM, Connolly RM, Moy B, Van Poznak CH, Blackwell KL, Puhalla SL, Jankowitz RC, Smith KL, Ibrahim N, Moynihan TJ, O'Sullivan CC, Nangia J, Niravath P, Tung N, Pohlmann PR, Burns R, Rimawi MF, Krop IE, Wolff AC, Winer EP, Lin NU; Translational Breast Cancer Research Consortium. TBCRC 022: A Phase II Trial of Neratinib and Capecitabine for Patients With Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer and Brain Metastases. J Clin Oncol. 2019 May 1;37(13):1081-1089. doi: 10.1200/JCO.18.01511. Epub 2019 Mar 12. PMID 30860945
- [Derived] Freedman RA, Gelman RS, Wefel JS, Melisko ME, Hess KR, Connolly RM, Van Poznak CH, Niravath PA, Puhalla SL, Ibrahim N, Blackwell KL, Moy B, Herold C, Liu MC, Lowe A, Agar NY, Ryabin N, Farooq S, Lawler E, Rimawi MF, Krop IE, Wolff AC, Winer EP, Lin NU. Translational Breast Cancer Research Consortium (TBCRC) 022: A Phase II Trial of Neratinib for Patients With Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer and Brain Metastases. J Clin Oncol. 2016 Mar 20;34(9):945-52. doi: 10.1200/JCO.2015.63.0343. Epub 2016 Feb 1. PMID 26834058

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patients With Progressive Brain Metastases. Intervention: HKI-272 (Neratinib) 240 mg orally, once daily.
- Cohort 2: Cohort 2 will be made up of participants who are candidates for craniotomy. They will be given Neratinib (240 mg orally daily).
- Cohort 3A: Cohort 3a will be made up of participants with No Prior Lapatinib Treatment. They will receive Neratinib 240mg Orally daily and 750mg/m2 Capecitabine twice per day for 14 days followed by 7 days rest.
- Cohort 3B: Cohort 3b will be made of participants with Prior Lapatinib Treatment. Cohort 3b participants will receive Neratinib 240mg Orally daily and 750mg/m2 Capecitabine twice per day for 14 days followed by 7 days rest.
- Cohort 4A: Cohort 4a will be made up of participants with previously untreated brain metastases. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
- Cohort 4B: Cohort 4b will be made up of participants with progressive brain metastases. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
- Cohort 4C: Cohort 4c will be made up of participants with progressive brain metastases and prior T-DM1. They will receive Neratinib 160mg Orally daily and T-DM1 3.6mg/kg IV every 3 weeks.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C
Started | 40 | 5 | 39 | 12 | 6 | 17 | 21
Completed | 40 | 5 | 37 | 12 | 6 | 17 | 21
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics reported for the subjects who completed the study, defined as all subjects who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C | Total
Number analyzed (Participants) | 40 | 5 | 37 | 12 | 6 | 17 | 21 | 138
Age, Continuous [Median (Full Range); unit: years] | 50 [34 to 69] | 43 [27 to 45] | 54 [31 to 64] | 52.5 [36 to 60] | 51 [43 to 65] | 48 [41 to 59] | 47 [34 to 67] | 50 [27 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 5 | 37 | 12 | 6 | 17 | 20 | 136
  Male | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 34 | 5 | 34 | 11 | 5 | 14 | 20 | 123
  Unknown or Not Reported | 3 | 0 | 2 | 0 | 0 | 3 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 34 | 5 | 32 | 7 | 4 | 14 | 20 | 116
  Race: Black or African American | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 7
  Race: Asian | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 5
  Race: Other or More than One Race | 2 | 0 | 2 | 3 | 1 | 2 | 0 | 10
Site of Metastatic Disease: Central Nervous System (CNS) Parenchymal [Count of Participants; unit: Participants]
  Yes | 40 | 5 | 37 | 12 | 6 | 17 | 21 | 138
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Site of Metastatic Disease: CNS Leptomeningeal [Count of Participants; unit: Participants]
  Yes | 4 | 1 | 2 | 1 | 0 | 1 | 2 | 11
  No | 36 | 4 | 35 | 11 | 6 | 16 | 19 | 127
  Unknown/Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Site of Metastatic Disease: Lung/Pleural [Count of Participants; unit: Participants]
  Yes | 15 | 0 | 9 | 4 | 1 | 3 | 6 | 38
  No | 25 | 5 | 28 | 8 | 5 | 14 | 15 | 100
Site of Metastatic Disease: Breast or Chest Wall [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 6 | 1 | 2 | 5 | 1 | 17
  No | 38 | 5 | 31 | 11 | 4 | 12 | 20 | 121
Site of Metastatic Disease: Lymph Node [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 6 | 2 | 1 | 2 | 6 | 17
  No | 40 | 5 | 31 | 10 | 5 | 15 | 15 | 121
Site of Metastatic Disease: Liver [Count of Participants; unit: Participants]
  Yes | 16 | 0 | 10 | 2 | 3 | 7 | 3 | 41
  No | 24 | 5 | 27 | 10 | 3 | 10 | 18 | 97
Site of Metastatic Disease: Bone [Count of Participants; unit: Participants]
  Yes | 26 | 0 | 21 | 2 | 5 | 9 | 13 | 76
  No | 14 | 5 | 16 | 10 | 1 | 8 | 8 | 62
Site of Metastatic Disease: Soft Tissue [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  No | 40 | 5 | 37 | 12 | 6 | 15 | 20 | 135
Estrogen Receptor Status (Metastatic Sample) [Count of Participants; unit: Participants]
  Negative | 18 | 4 | 16 | 6 | 1 | 7 | 11 | 63
  Positive | 22 | 0 | 21 | 6 | 5 | 8 | 7 | 69
  Missing | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 6
Has the patient had prior surgery for CNS tumors? [Count of Participants; unit: Participants]
  Yes | 12 | 3 | 11 | 3 | 0 | 7 | 7 | 43
  No | 28 | 2 | 26 | 9 | 6 | 10 | 14 | 95
Prior Stereotactic Radiosurgery (SRS) [Count of Participants; unit: Participants]
  Yes | 25 | 3 | 13 | 7 | 1 | 12 | 10 | 71
  No | 15 | 2 | 24 | 5 | 5 | 5 | 11 | 67
Prior Whole Brain Radiotherapy (WBRT) [Count of Participants; unit: Participants]
  Yes | 31 | 3 | 24 | 5 | 0 | 12 | 11 | 86
  No | 9 | 2 | 13 | 7 | 6 | 5 | 10 | 52

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Per Composite Response Criteria
Description: Defined as the percentage of patients achieving a complete response (CR) or partial response (PR) of Central Nervous System (CNS) lesions based on composite criteria, reported separately in Cohorts 1, 3A, 3B. For the volumetric criteria, an objective CR will be defined as the following: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks; no new lesions; stable or decreasing steroid dose; stable or improved neurological symptoms. An objective PR by volumetric criteria will be defined as the following: At least a 50% decrease in the sum volume of CNS target lesions, taking as reference the baseline sum volume sustained for at least 4 weeks; no new lesions; stable or decreasing steroid dose; stable or improved neurological symptoms.
Time Frame: 2 years
Population: ORR by composite criteria evaluated for all subjects who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Cohort 1: Patients With Progressive Brain Metastases. Intervention: HKI-272 (Neratinib)340 mg orally, once daily.
Arm/Group | Cohort 1 | Cohort 3A | Cohort 3B
Number analyzed (Participants) | 40 | 37 | 12
percent of participants | 7.5 [1.6 to 20.4] | 48.6 [31.9 to 65.6] | 33.3 [9.9 to 65.1]

2. Primary Outcome: Objective Response Rate Per RANO-BM Criteria
Description: Defined as the percentage of patients achieving a complete response (CR) or partial response (PR) of Central Nervous System (CNS) lesions based on RANO-BM criteria, reported separately in Cohorts 4A, 4B, and 4C. For the RANO-BM criteria, an objective CR will be defined as the following: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. An objective PR by RANO-BM criteria will be defined as the following: At least a 30% decrease in the sum LD of CNS target lesions, taking as reference the baseline sum LD sustained for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically.
Time Frame: 2 years
Population: Analysis population consists of all subjects who received at least one dose of treatment. All subjects enrolled in Cohorts 4A, 4B, and 4C received at least one dose of treatment, so all enrolled subjects are included in the objective response rate (ORR)
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 4A | Cohort 4B | Cohort 4C
Number analyzed (Participants) | 6 | 17 | 21
percent of participants | 33.3 [4.3 to 77.7] | 35.3 [14.2 to 61.7] | 28.6 [11.3 to 52.2]

3. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. A participant was considered to have an event if they had a CNS progression (defined by RANO-BM criteria for Cohort 4A, 4B, 4C, or defined by composite/volumetric criteria for Cohort 1 and Cohorts 3A and 3B), if they a non-CNS progression as defined by RECIST v1.1 criteria, or if they died without a progression within two cycle lengths (42 days) after their last scan date. Participants alive without disease progression are censored at the date of their last disease evaluation.
Time Frame: Assessed from date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
Population: PFS analyzed in all subjects who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C
Number analyzed (Participants) | 40 | 5 | 37 | 12 | 6 | 17 | 21
months | 1.9 [1.8 to 3.5] | 2.37 [2.07 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 5.5 [4.6 to 8.1] | 3.1 [1.97 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 5.26 [4.47 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 4.11 [2.69 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 4.14 [2.73 to 6.34]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the defined as the duration of time from the date of trial registration to death.
Time Frame: Assessed from date of trial registration until the date of death from any cause, up to 5 years
Population: OS evaluated for all subjects who completed the study, defined as all subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C
Number analyzed (Participants) | 40 | 5 | 37 | 12 | 6 | 17 | 21
months | 8.7 [4.9 to 15.1] | NA [6.24 to NA] — Both the median and the upper bound of confidence interval not estimable due to insufficient number of events | 13.3 [10.97 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 15.1 [7.0 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 30.16 [21.85 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 23.29 [17.64 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events | 20.86 [14.92 to NA] — Upper bound of confidence interval not estimable due to insufficient number of events

5. Secondary Outcome: CNS Response by Macdonald Criteria (Bidirectional Criteria)
Description: Defined as either a complete or partial response based on the Macdonald criteria. In the Macdonald response criteria, a complete response (CR) is defined as: disappearance of all enhancing tumor on consecutive CT or magnetic resonance imaging (MRI) scans at least 1 month apart, off steroids, and neurologically stable or improved. A partial response (PR) is defined as: at least 50% reduction in size of enhancing tumor on consecutive CT or MRI scans at least 1 month apart, steroids stable or reduced, and neurologically stable or improved. Reported for Cohort 1 only.
Time Frame: 2 years
Population: ORR by Macdonald (or bidirectional) criteria assessed for all subjects in Cohort 1 who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 40
percent of participants | 10.0 [2.8 to 23.7]

6. Secondary Outcome: Reason for Subject Being Taken Off Study Treatment
Description: Reason for subject being taken off study treatment: CNS progression, non-CNS progression, both CNS and non-CNS progression, or reason other than progression such as toxicity or physician decision. For subjects who came off treatment for progression, this outcome describes their first site of disease progression (CNS, non-CNS, or both).
Time Frame: 2 years
Population: Evaluated for all subjects who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C
Number analyzed (Participants) | 40 | 5 | 37 | 12 | 6 | 17 | 21
Participants
  CNS and Non-CNS Progression | 3 | 0 | 3 | 1 | 0 | 0 | 3
  CNS Progression | 29 | 2 | 23 | 8 | 3 | 11 | 12
  Non-CNS Progression | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Patient Withdrew for Other Reasons | 0 | 0 | 1 | 0 | 1 | 1 | 2
  Physician Discretion | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unacceptable Toxicity | 6 | 0 | 8 | 0 | 1 | 4 | 0
  Subject remained on study treatment at time of evaluation | 0 | 1 | 1 | 2 | 0 | 1 | 0
  Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Other off treatment reason | 0 | 2 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Objective Response Based on CNS Composite Criteria for Extension Subgroup of Cohort 1
Description: Assess number of objective responses based on CNS composite criteria for subjects in Cohort 1 who opt to receive trastuzumab and neratinib at the time of non-CNS progression
Time Frame: 2 years
Population: Of the total 40 subjects in Cohort 1, two patients who experienced non-CNS progression received trastuzumab-neratinib on the extension cohort after one and two cycles of neratinib, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Objective Response Rate in CNS by Volumetric Criteria
Description: Defined as the percentage of patients achieving a complete response (CR) or partial response (PR) of Central Nervous System (CNS) lesions based on volumetric criteria, reported separately in Cohorts 4A, 4B, and 4C. For the volumetric criteria, an objective CR will be defined as the following: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks; no new lesions. An objective PR by volumetric criteria will be defined as the following: At least a 50% decrease in the sum volume of CNS target lesions, taking as reference the baseline sum volume sustained for at least 4 weeks; no new lesions.
Time Frame: 2 years
Population: Objective response rate in CNS by volumetric criteria evaluated for all subjects who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 4A | Cohort 4B | Cohort 4C
Number analyzed (Participants) | 6 | 17 | 21
percent of participants | 50.0 [11.8 to 88.2] | 29.4 [10.3 to 56.0] | 23.8 [8.2 to 47.2]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 5 years; all adverse events were collected up to 4 years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 4C
All-Cause Mortality (participants affected / at risk) | 34/40 | 2/5 | 21/37 | 6/12 | 3/6 | 8/17 | 11/21
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/5 | 0/37 | 0/12 | 0/6 | 1/17 | 0/21
Other Adverse Events (participants affected / at risk) | 38/40 | 5/5 | 35/37 | 12/12 | 6/6 | 17/17 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=40) | Cohort 2 (N=5) | Cohort 3A (N=37) | Cohort 3B (N=12) | Cohort 4A (N=6) | Cohort 4B (N=17) | Cohort 4C (N=21)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=40) | Cohort 2 (N=5) | Cohort 3A (N=37) | Cohort 3B (N=12) | Cohort 4A (N=6) | Cohort 4B (N=17) | Cohort 4C (N=21)
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 2 | 2 | 2 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1 | 2 | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1 | 2 | 1 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 1 | 2 | 1 | 1 | 3 | 1
Dry eye (Eye disorders) | 1 | 2 | 1 | 2 | 1 | 1 | 1
Photophobia (Eye disorders) | 1 | 2 | 2 | 1 | 1 | 1 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 2 | 2 | 1 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 5 | 1 | 1 | 5
Bloating (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 1 | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 11 | 6 | 10 | 1
Constipation (Gastrointestinal disorders) | 13 | 1 | 8 | 1 | 1 | 13 | 16
Diarrhea (Gastrointestinal disorders) | 32 | 1 | 32 | 8 | 1 | 4 | 17
Dry mouth (Gastrointestinal disorders) | 5 | 1 | 1 | 5 | 2 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 2 | 5 | 3 | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 3 | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 3 | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 5 | 3 | 1 | 11
Oral pain (Gastrointestinal disorders) | 2 | 1 | 5 | 5 | 3 | 1 | 1
Stomach pain (Gastrointestinal disorders) | 5 | 1 | 1 | 5 | 3 | 2 | 1
Vomiting (Gastrointestinal disorders) | 13 | 1 | 5 | 5 | 3 | 11 | 9
Vomiting (Gastrointestinal disorders) | 8 | 1 | 23 | 5 | 3 | 9 | 9
Oral pain (Gastrointestinal disorders) | 8 | 1 | 1 | 5 | 3 | 9 | 9
Vomiting (Gastrointestinal disorders) | 8 | 1 | 21 | 5 | 3 | 9 | 9
Fatigue (General disorders) | 20 | 2 | 2 | 1 | 4 | 1 | 9
General disorders and administration site conditions - Other, specify (General disorders) | 3 | 2 | 1 | 4 | 1 | 8 | 1
Non-cardiac chest pain (General disorders) | 1 | 2 | 19 | 3 | 1 | 1 | 1
Pain (General disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 2
Infusion related reaction (General disorders) | 1 | 2 | 3 | 1 | 1 | 1 | 2
Infusion site extravasation (General disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 2
Pain (General disorders) | 1 | 2 | 5 | 1 | 1 | 1 | 2
Edema face (General disorders and administration site conditions) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders and administration site conditions) | 7 | 0 | 19 | 1 | 0 | 0 | 0
Fatigue (General disorders and administration site conditions) | 20 | 0 | 19 | 1 | 0 | 0 | 0
Gait disturbance (General disorders and administration site conditions) | 1 | 0 | 19 | 1 | 0 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 3 | 0 | 19 | 1 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 1
Papulopustular rash (Infections and infestations) | 2 | 1 | 2 | 0 | 1 | 1 | 1
Paronychia (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 1 | 1
Rhinitis infective (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 3 | 2 | 0 | 1 | 2 | 1
Upper respiratory infection (Infections and infestations) | 2 | 3 | 3 | 0 | 1 | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1 | 5 | 2 | 2 | 5 | 5
Alkaline phosphatase increased (Investigations) | 1 | 1 | 4 | 2 | 2 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 3 | 6 | 6
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 1 | 2 | 1 | 2
Platelet count decreased (Investigations) | 1 | 1 | 1 | 1 | 1 | 1 | 5
Weight loss (Investigations) | 1 | 1 | 1 | 1 | 1 | 3 | 1
White blood cell decreased (Investigations) | 1 | 1 | 2 | 1 | 1 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 9 | 1 | 10 | 2 | 1 | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 3 | 3 | 1 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 1 | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 6 | 1 | 1 | 1 | 1 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 1 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 5 | 1 | 1 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 1 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 1 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 0 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4 | 0 | 4 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 4 | 0 | 1 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 4 | 0 | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 3 | 1 | 1 | 1 | 1 | 2 | 1
Encephalopathy (Nervous system disorders) | 9 | 1 | 1 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 4 | 5 | 1 | 2 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1 | 2 | 1 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 8 | 1 | 1 | 1 | 2
Seizure (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 8 | 3
Intracranial hemorrhage (Nervous system disorders) | 9 | 1 | 10 | 1 | 1 | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 1 | 1 | 1 | 2 | 3
Tremor (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 3
Seizure (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 3
Syncope (Nervous system disorders) | 6 | 1 | 1 | 1 | 1 | 2 | 3
Syncope (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 4 | 1 | 1 | 1 | 1 | 1 | 2
Depression (Psychiatric disorders) | 1 | 1 | 3 | 1 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 5 | 1 | 1 | 2 | 1 | 1 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1 | 1 | 3 | 8
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 1 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 3 | 2 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 4
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 10 | 1 | 2 | 2 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 1 | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 6 | 1 | 2 | 1 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 1 | 2 | 1 | 1
Lymphedema (Vascular disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT01494662/Prot_SAP_000.pdf